CLINICAL TRIAL: NCT01269801
Title: A Phase IV Prospective, Open Label, Randomized, Crossover Study Evaluating BOTOX Cosmetic for Injection and JUVEDERM Injectable Gel for the Treatment of Moderate to Severe Facial Wrinkles and Folds
Brief Title: Study of BOTOX and JUVEDERM for Treatment of Moderate to Severe Facial Wrinkles and Folds
Acronym: JUVE_BTX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AboutSkin Dermatology and DermSurgery, PC (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, AboutSkin Dermatology, Joel L. Cohen, MD, AboutSkin Dermatology and DermSurgery, PC
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JUVE_BTX-09-01
Record Dates: First submitted 2011-01-02; First posted 2011-01-04 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Wrinkles
Keywords: BOTOX; JUVEDERM; Prospective; Open Label; Randomized; Crossover Study
MeSH Terms: interventions — Botulinum Toxins, Type A; WW Domain-Containing Oxidoreductase; Juvéderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox Cosmetic (Active Comparator): onabotulinumtoxinA for injection
  Interventions: Drug: onabotulinumtoxinA
- JUVÉDERM (Active Comparator): JUVÉDERM® Ultra XC and JUVÉDERM® Ultra Plus XC Injectable Gel
  Interventions: Drug: JUVÉDERM

INTERVENTIONS:
Drug: onabotulinumtoxinA — * Group 1 will initially receive BOTOX® Cosmetic or VISTABEL® injections to the affected facial regions;
  * Group 2 will initially receive JUVÉDERM® Ultra XC or JUVÉDERM® Ultra 2 (for moderate facial lines or folds) or JUVÉDERM® Ultra Plus XC or JUVÉDERM® Ultra 3 (for severe facial lines or folds) injections to the affected facial regions.
  At 4 weeks,Group 1 patients who initially received BOTOX® Cosmetic or VISTABEL® treatment will be crossed over and receive JUVÉDERM® treatment, and Group 2 patients who initially received JUVÉDERM® treatment will be crossed over to receive BOTOX® Cosmetic or VISTABEL® treatment.
  Other Names: Europe Investigative Sites:; VISTABEL® (Botulinum toxin type A) for Injection
  Arms: Botox Cosmetic
Drug: JUVÉDERM — Group 1 will initially receive BOTOX® Cosmetic or VISTABEL® injections to the affected facial regions;
  • Group 2 will initially receive JUVÉDERM® Ultra XC or JUVÉDERM® Ultra 2 (for moderate facial lines or folds) or JUVÉDERM® Ultra Plus XC or JUVÉDERM® Ultra 3 (for severe facial lines or folds) injections to the affected facial regions.
  At 4 weeks,Group 1 patients who initially received BOTOX® Cosmetic or VISTABEL® treatment will be crossed over and receive JUVÉDERM® treatment, and Group 2 patients who initially received JUVÉDERM® treatment will be crossed over to receive BOTOX® Cosmetic or VISTABEL® treatment.
  Other Names: EU Investigative Sites:; JUVÉDERM® Ultra 2 and JUVÉDERM® Ultra 3 Injectable Gel
  Arms: JUVÉDERM

SUMMARY:
The purpose of this study is to see how well Juvederm Ultra XC or Juvederm Ultra Plus XC, and BOTOX Cosmetic, work compared to each other and when used together for the cosmetic treatment of age-associated wrinkles and folds of the face.

DETAILED DESCRIPTION:
1. Compounds:

   1. BOTOX Cosmetic (onabotulinumtoxinA) for Injection
   2. JUVEDERM Ultra XC and JUVEDERM Ultra Plus XC Injectable Gel
2. The objectives of this study are:

   1. To assess physician assessment of efficacy and incremental benefit following BOTOX Cosmetic and Juvederm for the treatment of moderate to severe facial wrinkles and folds;
   2. To assess patient perceptions of treatment outcomes and incremental benefit following BOTOX Cosmetic and Juvederm for the treatment of moderate to severe facial wrinkles and folds.
3. Investigator and study sites:

   1. multicenter study
   2. 5 Sites: 2 in US, 2 in Canada, 1 in EU

ELIGIBILITY:
Inclusion Criteria:

* Adult females or males, aged 25 to 65 years;
* Subjects must be seeking treatment with either BOTOX® or JUVÉDERM injections;
* Subjects must have one or more moderate to severe hyperfunctional facial lines of the upper face (i.e., glabellar lines, lateral canthal lines (crow's feet) or horizontal forehead lines) or moderate to severe nasolabial folds based on the physician observer assessment (0-3 scale);
* Women must either be of non-childbearing potential (i.e., surgically sterilized or post-menopausal) or if of childbearing potential, must not be pregnant (as documented by a negative urine pregnancy test at the baseline examination) or lactating and must be practicing a medically acceptable method of birth control;
* Subjects must be willing and able to provide written informed consent;
* Subjects must be willing and able to follow the procedures outlined in this protocol.

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test) or who have an infant they are breast-feeding or who are of childbearing potential and not practicing a reliable method of birth control;
* Previous botulinum toxin or semipermanent injectable filler therapy within the past year or any prior history of permanent filler therapy injection;
* Prior cosmetic procedures (i.e., liposuction, etc.) or visible scars that may affect evaluation of response and/or quality of photography;
* Known allergy or sensitivity to any of the study medication or their components;
* Known severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies;
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis or any other disease that might interfere with neuromuscular function;
* Concurrent use of aminoglycoside antibiotics that interfere with neuromuscular function;
* Subjects with profound atrophy or excessive weakness of the muscles in the target area(s) of BOTOX injection;
* Subjects with an infection at an injection site or systemic infection (in this case, postpone study entry until one week following recovery);
* Concurrent participation in an investigational drug or device study or participation within 30 days of study start;
* Subjects are not to undergo any additional cosmetic procedures during the study period;
* Subjects are not to change use of any facial products up to 6 months prior to enrollment and during study period;
* Subjects with a history of poor cooperation, non-compliance with medical treatment, or unreliability.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel L Cohen, MD, Principal Investigator — AboutSkin Dermatology and DermSurgery, PC
Locations (3):
- About Skin Dermatology, Englewood, Colorado, United States
- Canada (2):
  - Niagara Falls Dermantology and Skin Care Center, Niagara Falls, Ontario
  - University of Toronto, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized to two groups: Juvederm first, then Botox (Juvederm group) or Botox first, then Juvederm (Botox group).
  For the Juvederm group, Day 1 involved juvederm treatment. Week 4 involved botox administration.
  For the Botox group, Day 1 involved botox treatment. Week 4 involved juvederm administration.
Groups:
- JUVÉDERM: JUVÉDERM® Ultra XC and JUVÉDERM® Ultra Plus XC Injectable Gel
  Juvederm group will initially receive JUVÉDERM® Ultra Plus XC or JUVÉDERM® Ultra 3 (for severe facial lines or folds) injections to the affected facial regions at Day 1.
  At Week 4, patients who initially received JUVÉDERM® treatment will be crossed over to receive BOTOX® Cosmetic or VISTABEL® treatment.
- Botox Cosmetic: Botox group will initially receive BOTOX® Cosmetic injections to the affected facial regions at Day 1.
  At Week 4, patients who initially received BOTOX® Cosmetic treatment will be crossed over to receive JUVÉDERM® Ultra XC and JUVÉDERM® Ultra Plus XC Injectable Gel treatment.
Period: Overall Study
Arm/Group | JUVÉDERM | Botox Cosmetic
Started | 74 | 80
Completed | 74 | 77
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis stratified by treatment group (per sequence).
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox Cosmetic | JUVÉDERM | Total
Number analyzed (Participants) | 80 | 74 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 74 | 154
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.83 (7.42) | 51.12 (7.78) | 50.54 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 66 | 142
  Male | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Efficacy
Description: Assessments at Visits 3,5,6+7 (weeks 4,8,12,24) include:
  -Physician Global Aesthetic Improvement Scale (PGAIS). Ratings include no change, improved, much improved, very much improved.
  Number of subjects with improvement score for the 5 point PGAIS from baseline to Visit 7.
  -Objective Observer Global Aesthetic Improvement Scale Number of subjects with improvement score for the from baseline to Visit 7. Ratings include no change, some improvement, definite improvement, substantial improvement, and complete improvement.
Time Frame: Week 4, 8, 12, 24
Population: Analysis is based on the randomization group to account for the order in which the products were administered.
Measure: Number; unit: participantes rated improved and higher
Arm/Group | Botox Cosmetic | JUVÉDERM
Number analyzed (Participants) | 77 | 74
participantes rated improved and higher
  PGAIS Week 24 | 77 | 74
  Objective Observer global assessment Week 24 | 73 | 72
  PGAIS Week 12 | 77 | 74
  Objective Observer global assessment Week 12 | 77 | 74
  PGAIS Week 8 | 78 | 73
  Objective Observer global assessment Week 8 | 78 | 73
  PGAIS Week 4 | 75 | 74
  Objective Observer global assessment Week 4 | 72 | 74

ADVERSE EVENTS:
Time Frame: Week 4, 8, 12, 24
Description: Adverse Events assessed based on treatment received before the adverse event onset.
Arm/Group | Botox Cosmetic | JUVÉDERM
Serious Adverse Events (participants affected / at risk) | 1/154 | 0/152
Other Adverse Events (participants affected / at risk) | 8/154 | 19/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox Cosmetic (N=154) | JUVÉDERM (N=152)
death due to hypertensive cardiovascular disease (Vascular disorders) | 1 (1) | 0 (0) — Subject died 2 months after last study visit, approximately 1.5 months after last juvederm injection. Investigator assessed as not related to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox Cosmetic (N=154) | JUVÉDERM (N=152)
(Contusion) Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 19 (19)
Facial Paresis (Nervous system disorders) | 8 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No